CLINICAL TRIAL: NCT06373770
Title: Effects of Ayres Sensory Integration Therapy Versus Conservative Treatment in Autism Spectrum
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MSRSW/Batch-Fall22/700
Record Dates: First submitted 2024-04-16; First posted 2024-04-18 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ayres sensory integration therapy (Experimental): A. Jean Ayres, is a theory and practice that targets a person's ability to process and internally integrate sensory information from their body and environment.
  Interventions: Diagnostic Test: Ayres sensory integration therapy
- Behaviour therapy (Other): The current treatment options for the core symptoms of autism are limited to psychosocial therapies, such as applied behavior analysis.
  Interventions: Diagnostic Test: Behaviour Therapy

INTERVENTIONS:
Diagnostic Test: Ayres sensory integration therapy — A. Jean Ayres, is a theory and practice that targets a person's ability to process and internally integrate sensory information from their body and environment. Sensory information may be visual, auditory, tactile, proprioceptive, and/or vestibular in nature. ASI uses individually tailored activities that utilize "just right" challenges to an individual's existing patterns of sensory processing and motor planning and encourage movement and organization of self in time and space. ASI incorporates specialized equipment and materials in purposeful and playful activities in order to improve adaptive behavior.
  Arms: Ayres sensory integration therapy
Diagnostic Test: Behaviour Therapy — The current treatment options for the core symptoms of autism are limited to psychosocial therapies, such as applied behavior analysis. Medications have been most effective in treating the associated behavioral symptoms of autism, though studies have examined potential benefits in some of the core symptoms of autism with certain medications, especially the repetitive behaviors often seen with this diagnosis. Risperidone and aripiprazole are currently the only medications FDA approved for symptoms associated with autism spectrum disorders, targeting the irritability often seen with this diagnosis.
  Arms: Behaviour therapy

SUMMARY:
Effects of Ayres Sensory Integration Therapy Versus Conservative Treatment in Autism Spectrum

DETAILED DESCRIPTION:
"This study named effects of ayres sensory integration therapy versus conservative treatment in autism spectrum is a randomized clinical trail study.There is no evidence-based intervention protocol to treat sensory integration dysfunction in autism spectrum. This study may help finding best therapeutic treatment approach for sensory integration dysfunction results in repetitive behavior and impairments in functionality in autism spectrum.This study helps

* To evaluate best intervention plan for sensory integration dysfunction, Ayres sensory integration therapy versus conservative treatment in autism spectrum.
* To determine how many patients will be having what type of sensory integration dysfunction that come with autism spectrum leading to certain level of functional restrictions in Activity of Daily Livings (ADLs).
* Which type of sensory integration dysfunction having greater functional impairment and need to be focused more for intervention?
* To make better individualized rehabilitation treatment plan being an Occupational Therapist."

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases of autism age range from 2 year to 8 years.
* All patients will be assed using sensory profile by Winnie Dunn.
* All the patients fulfilling the above-mentioned inclusion criteria will be assessed and evaluated by occupational therapist for sensory integration dysfunction.

Exclusion Criteria:

* All other patients not having diagnosed as autism spectrum criteria are excluded.
* All patients with sensory processing disorder assessed by using sensory profile.

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
sensory profile by winnie dunn | 12 Months
  sensory profile by winnie dunn willl be used to measure primary outcomes or initial assessment

CONTACTS AND LOCATIONS:
Locations (1):
- RICCER Institute, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No